CLINICAL TRIAL: NCT00546572
Title: A Phase 3, Randomized, Active-Controlled, Modified Double-Blind Trial, Evaluating The Safety, Tolerability And Immunogenicity Of A 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) Compared To A 23-Valent Pneumococcal Polysaccharide (23vPS) Vaccine in Ambulatory Elderly Individuals Aged 70 Years And Older Who Received One Dose of 23vPS At Least 5 Years Prior To Study Enrollment
Brief Title: Study Evaluating The Safety, Tolerability And Immunogenicity Of A 13-Valent Pneumococcal Conjugate Vaccine (13vPnC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6115A1-3005; B1851024
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Results first posted 2011-05-30 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receives 13vPnC at year 0 and 13vPnC at year 1
  Interventions: Biological: 13 valent Pneumococcal Conjugate Vaccine
- 2 (Active Comparator): Receives 23vPS at year 0 and 13vPnC at year 1
  Interventions: Biological: 23vPS

INTERVENTIONS:
Biological: 13 valent Pneumococcal Conjugate Vaccine — 0.5-mL dose 13vPnC will be administered into the deltoid muscle at year 0 and year 1
  Arms: 1
Biological: 23vPS — 0.5-mL dose 23vPS will be administered into the deltoid muscle at year 0 and 0.5-mL dose 13vPnC will be administered into the deltoid muscle at year 1
  Arms: 2

SUMMARY:
This study will evaluate the safety, tolerability and immunogenicity of study vaccines 13vPnC and 23vPS in older, healthy subjects who have previously received a dose of 23vPS at least 5 years ago. It will also evaluate the safety, tolerability and immunogenicity to a dose of 13vPnC 1 year after the initial dose of study vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 70 years or older.
* Documented vaccination with 1 dose of 23vPS at least 5 years previous.
* Healthy.

Exclusion Criteria:

* Receipt of more than one dose of 23vPS prior to enrollment.
* History of severe adverse reaction to a vaccine.
* Immunodeficiency.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 938 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (46):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Stockbridge, Georgia
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Corvallis, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Carnegie, Pennsylvania
  - Pfizer Investigational Site, Downington, Pennsylvania
  - Pfizer Investigational Site, Grove City, Pennsylvania
  - Pfizer Investigational Site, Penndel, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Upper Saint Clair, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Sweden (7):
  - Pfizer Investigational Site, Arlöv
  - Pfizer Investigational Site, Boden
  - Pfizer Investigational Site, Degeberga
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Uppsala

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3005&StudyName=Study%20Evaluating%20The%20Safety%2C%20Tolerability%20And%20Immunogenicity%20Of%20A%2013-Valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC / 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliters (mL) dose intramuscularly (IM) at Year 0 (vaccination 1 [Vax 1]) and 13vPnC 0.5 mL IM at Year 1 (Vax 2)
- 23vPS / 13vPnC: 23-valent pneumococcal polysaccharide conjugate vaccine (23vPS) 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL IM at Year 1 (Vax 2)
Period: Vax 1 / Year 0
Arm/Group | 13vPnC / 13vPnC | 23vPS / 13vPnC
Started | 464 | 474
Received Vax 1 | 463 | 473
Completed | 391 | 404
Not Completed | 73 | 70
Not completed — Randomized, not treated | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 3 | 4
Not completed — Death | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — 6-Month Contact; withdraw before Vax 2 | 64 | 59
Period: Vax 2 / Year 1
Arm/Group | 13vPnC / 13vPnC | 23vPS / 13vPnC
Started | 391 | 404
Received Vax 2 | 391 | 404
Completed | 387 | 402
Not Completed | 4 | 2
Not completed — Other | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Vax 2; withdraw before 6-Month Contact | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC: 13vPnC 0.5 mL dose IM at Year 0 (Vax 1)
- 23vPS: 23vPS 0.5 mL dose IM at Year 0 (Vax 1)
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 23vPS | Total
Number analyzed (Participants) | 463 | 473 | 936
Age Continuous [Mean (Standard Deviation); unit: years] | 76.7 (4.6) | 76.7 (4.5) | 76.7 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 235 | 456
  Male | 242 | 238 | 480

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 13vPnC Relative to 23vPS (Vax 1 / Year 0)
Description: Antibody geometric mean titers as measured by opsonophagocytic activity (OPA) assays for the 12 common serotypes (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after Vax 1 / Year 0
Population: Evaluable Immunogenicity population: treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations. N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 426 | 445
geometric mean titer
  Serotype 1 | 81 [68.4 to 95.9] | 55 [46.2 to 64.8]
  Serotype 3 | 55 [47.7 to 62.9] | 49 [42.9 to 56.9]
  Serotype 4 | 545 [441.9 to 672.3] | 203 [157.1 to 262.2]
  Serotype 5 | 72 [59.7 to 86.6] | 36 [29.5 to 43.1]
  Serotype 6B | 1261 [1024.7 to 1552.6] | 417 [330.5 to 526.7]
  Serotype 7F | 245 [191.9 to 312.4] | 160 [123.5 to 207.9]
  Serotype 9V | 181 [138.0 to 237.0] | 90 [67.8 to 119.7]
  Serotype 14 | 280 [227.5 to 345.5] | 285 [228.9 to 354.3]
  Serotype 18C | 907 [761.9 to 1080.1] | 481 [385.1 to 600.7]
  Serotype 19A | 354 [307.7 to 408.4] | 200 [170.0 to 234.4]
  Serotype 19F | 333 [273.2 to 404.8] | 214 [174.3 to 262.8]
  Serotype 23F | 158 [126.0 to 198.6] | 43 [34.2 to 53.5]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Serotype 1: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — Non-inferiority declared if the lower limit of the 2-sided 95 % confidence interval for the geometric mean ratio (GMR) was > 0.5 (2-fold criterion). Statistical significance demonstrated if the lower limit of the 2-sided 95 % confidence interval for the geometric mean ratio (GMR) was > 1; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.17 to 1.88] — Confidence intervals for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS)
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS; Serotype 3: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.1, 95% CI 2-sided [0.91 to 1.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 23vPS; Serotype 4: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.7, 95% CI 2-sided [1.93 to 3.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 23vPS; Serotype 5: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.0, 95% CI 2-sided [1.55 to 2.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 23vPS; Serotype 6B: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 3.0, 95% CI 2-sided [2.21 to 4.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 23vPS; Serotype 7F: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.07 to 2.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 23vPS; Serotype 9V: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. Statistical significance demonstrated if the lower limit of the 2-sided 95 % confidence interval for the geometric mean ratio (GMR) was > 1; Test type: Non-Inferiority or Equivalence — Non-inferiority declared if the lower limit of the 2-sided 95 % confidence interval for the geometric mean ratio (GMR) was > 0.5 (2-fold criterion); ratio of geometric mean titer = 2.0, 95% CI 2-sided [1.36 to 2.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 23vPS; Serotype 14: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.0, 95% CI 2-sided [0.73 to 1.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 23vPS; Serotype 18C: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.9, 95% CI 2-sided [1.42 to 2.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 23vPS; Serotype 19A: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.8, 95% CI 2-sided [1.43 to 2.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 23vPS; Serotype 19F: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.17 to 2.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 23vPS; Serotype 23F: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 3.7, 95% CI 2-sided [2.69 to 5.09] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Achieving a ≥ 4-fold Rise for Serotype 6A OPA Titer for 13vPnC Relative to 23vPS (Vax 1 / Year 0)
Description: OPA titer for the 6A serotype measured for at least a 4-fold increase from the prevaccination to postvaccination blood sample collection. Exact 2-sided CI (Clopper and Pearson) based upon the observed percentage of participants.
Time Frame: Baseline, 1 month after Vax 1 / Year 0
Population: Evaluable Immunogenicity population. N=number of participants with a determinate antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 408 | 411
observed percentage of participants | 71.1 [66.4 to 75.4] | 27.3 [23.0 to 31.8]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Serotype 6A: difference in proportions, 13vPnC - 23vPS, expressed as a percentage. Statistical significance was shown if the lower limit of the 95% CI for the difference in proportions (13vPnC - 23vPS) was > 0; Test type: Superiority or Other; difference in proportions = 43.8, 95% CI 2-sided [37.4 to 49.9] — Exact 2-sided CI (based on Chan and Zhang) for the difference in proportions, 13vPnC - 23vPS expressed as a percentage

3. Secondary Outcome: Pneumococcal OPA Geometric Mean Titer (GMT) for Serotype 6A for 13vPnC Relative to 23vPS (Vax 1 / Year 0)
Description: Antibody geometric mean titer as measured by OPA assay for the 6A pneumococcal serotype. Confidence intervals for the GMT are back transformation of a CI based on the Student t distribution for the mean logarithm of the titer.
Time Frame: 1 month after Vax 1 / Year 0
Population: Evaluable Immunogenicity population. N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 421 | 433
geometric mean titer | 903 [726.7 to 1121.3] | 94 [74.1 to 118.5]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Serotype 6A: ratio of GMT (13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. Statistical significance was demonstrated if the lower limit of the 2-sided 95% confidence interval for the geometric mean ratio was >2; Test type: Superiority or Other; ratio of geometric mean titer = 9.6, 95% CI 2-sided [7.00 to 13.26] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 13 Serotypes for 13vPnC / 13vPnC (Vax 2 / Year 1) Relative to 13vPnC (Vax 1 / Year 0)
Description: Antibody geometric mean titers as measured by OPA assays for the 13 serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after Vax 1 / Year 0, 1 month after Vax 2 / Year 1
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the given serotype at both the postvaccination 1 and postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC / 13vPnC: 13vPnC 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax 2)
Arm/Group | 13vPnC | 13vPnC / 13vPnC
Number analyzed (Participants) | 361 | 361
geometric mean titer
  Serotype 1 | 79 [65.3 to 94.6] | 76 [64.8 to 89.7]
  Serotype 3 | 55 [47.2 to 64.0] | 55 [48.4 to 63.1]
  Serotype 4 | 614 [489.8 to 768.8] | 487 [393.9 to 603.3]
  Serotype 5 | 69 [56.2 to 84.2] | 57 [46.9 to 68.5]
  Serotype 6A | 971 [771.0 to 1222.1] | 1169 [974.0 to 1403.0]
  Serotype 6B | 1358 [1085.4 to 1700.2] | 1590 [1316.9 to 1919.8]
  Serotype 7F | 222 [170.2 to 290.2] | 180 [138.1 to 233.8]
  Serotype 9V | 187 [139.3 to 250.4] | 166 [124.2 to 220.8]
  Serotype 14 | 265 [209.9 to 333.6] | 241 [194.4 to 299.1]
  Serotype 18C | 918 [763.4 to 1104.3] | 1003 [850.2 to 1182.1]
  Serotype 19A | 349 [299.7 to 405.5] | 341 [297.2 to 390.5]
  Serotype 19F | 329 [265.6 to 408.6] | 322 [266.3 to 389.6]
  Serotype 23F | 167 [130.9 to 213.0] | 309 [251.6 to 380.1]
Statistical Analysis 1: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 1: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — Non-inferiority declared if the lower limit of the 95% confidence interval for the back-transformed GMFR was > 0.5 (2-fold criterion); geometric mean fold rise = 1.0, 95% CI 2-sided [0.85 to 1.10] — Confidence intervals are back transformations of a CI based on the student t distribution for the mean logarithm of the titers
Statistical Analysis 2: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 3: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.0, 95% CI 2-sided [0.91 to 1.11] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 4: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.68 to 0.92] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 5: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.73 to 0.94] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 6A: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.2, 95% CI 2-sided [1.03 to 1.40] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 6B: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.2, 95% CI 2-sided [1.02 to 1.35] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 7F: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.65 to 1.01] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 9V: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 0.9, 95% CI 2-sided [0.69 to 1.15] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 14: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 0.9, 95% CI 2-sided [0.79 to 1.05] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 18C: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.1, 95% CI 2-sided [0.97 to 1.23] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 19A: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.0, 95% CI 2-sided [0.89 to 1.07] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 19F: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.0, 95% CI 2-sided [0.83 to 1.15] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 13vPnC / 13vPnC; Serotype 23F: geometric mean fold rise (GMFR) [(13vPnC / 13vPnC) / (13vPnC)] calculated using all participants with available data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean fold rise = 1.9, 95% CI 2-sided [1.60 to 2.14] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 13vPnC / 13vPnC (Vax 2 / Year 1) Relative to 23vPS (Vax 1 / Year 0)
Description: Antibody geometric mean titers as measured by OPA assays for the 12 common serotypes (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after Vax 1 / Year 0, 1 month after Vax 2 / Year 1
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titers
Arm/Group | 13vPnC / 13vPnC | 23vPS
Number analyzed (Participants) | 370 | 445
geometric mean titers
  Serotype 1 | 76 [64.9 to 89.5] | 55 [46.2 to 64.8]
  Serotype 3 | 55 [47.9 to 62.0] | 49 [42.9 to 56.9]
  Serotype 4 | 472 [383.5 to 580.2] | 203 [157.1 to 262.2]
  Serotype 5 | 56 [46.6 to 67.7] | 36 [29.5 to 43.1]
  Serotype 6B | 1565 [1306.1 to 1875.9] | 417 [330.5 to 526.7]
  Serotype 7F | 185 [142.9 to 239.7] | 160 [123.5 to 207.9]
  Serotype 9V | 158 [119.5 to 209.5] | 90 [67.8 to 119.7]
  Serotype 14 | 238 [192.3 to 293.8] | 285 [228.9 to 354.3]
  Serotype 18C | 975 [829.0 to 1147.3] | 481 [385.1 to 600.7]
  Serotype 19A | 339 [296.4 to 386.9] | 200 [170.0 to 234.4]
  Serotype 19F | 311 [257.1 to 375.9] | 214 [174.3 to 262.8]
  Serotype 23F | 310 [254.1 to 378.0] | 43 [34.2 to 53.5]
Statistical Analysis 1: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 1: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.4, 95% CI 2-sided [1.10 to 1.76] — Confidence intervals for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(13vPnC / 13vPnC )- (23vPS)]
Statistical Analysis 2: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 3: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.1, 95% CI 2-sided [0.91 to 1.34] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 4: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 2.3, 95% CI 2-sided [1.66 to 3.25] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 5: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.21 to 2.06] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 6B: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 3.8, 95% CI 2-sided [2.78 to 5.07] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 7F: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.2, 95% CI 2-sided [0.80 to 1.67] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 9V: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.8, 95% CI 2-sided [1.18 to 2.62] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 14: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 0.8, 95% CI 2-sided [0.62 to 1.13] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 18C: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 2.0, 95% CI 2-sided [1.53 to 2.69] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 19A: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.7, 95% CI 2-sided [1.37 to 2.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 19F: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.09 to 1.93] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 23F: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 7]; ratio of geometric mean titer = 7.3, 95% CI 2-sided [5.36 to 9.82] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Pneumococcal OPA Geometric Mean Titer (GMT) for Serotype 6A for 13vPnC / 13vPnC (Vax 2 / Year 1) Relative to 23vPS (Vax 1 / Year 0)
Description: Antibody geometric mean titer as measured by OPA assay for the 6A serotype. Confidence intervals (CI) for the GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titer.
Time Frame: 1 month after Vax 1 / Year 0, 1 month after Vax 2 / Year 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | 13vPnC / 13vPnC | 23vPS
Number analyzed (Participants) | 366 | 433
geometric mean titer | 1134 [943.6 to 1363.7] | 94 [74.1 to 118.5]
Statistical Analysis 1: Comparison: 13vPnC / 13vPnC vs 23vPS; Serotype 6A: ratio of GMT (13vPnC / 13vPnC to 23vPS) calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. Statistical significance was demonstrated if the lower limit of the 2-sided 95% confidence interval for the geometric mean ratio was >2; Test type: Superiority or Other; ratio of geometric mean titer = 12.1, 95% CI 2-sided [8.92 to 16.44] — [estimate comment as in outcome 5, analysis 1]

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for 13vPnC and 23vPS (Vax 1 / Year 0)
Description: Local reactions reported in electronic diary. Redness and swelling scaled as Any (redness or swelling present); Mild (2.5 centimeters [cm] to 5.0 cm); Moderate (5.1 to 10.0 cm); Severe (>10.0 cm). Pain scaled as Any (pain present); Mild (awareness of symptom, easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating, inability to do usual activity). Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move above head, able to move above shoulder); Severe (unable to move above shoulder)
Time Frame: Days 1 through 14 / Year 0
Population: Safety population is all participants who receive at least 1 dose of study vaccine. N=number of participants who reported any local reaction reactogenicity events; (n)=number of participants with known values for 13vPnC and 23vPS (Vax 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 370 | 387
percentage of participants
  Redness: Any (n=306, 324) | 10.8 | 22.2
  Redness: Mild (n=304, 311) | 9.5 | 13.5
  Redness: Moderate (n=301, 314) | 4.7 | 11.5
  Redness: Severe (n=299, 310) | 1.7 | 4.8
  Swelling: Any (n=307, 333) | 10.4 | 23.1
  Swelling: Mild (n=305, 315) | 8.9 | 14.0
  Swelling: Moderate (n=299, 323) | 4.0 | 13.6
  Swelling: Severe (n=297, 310) | 0.0 | 4.8
  Pain: Any (n=362, 383) | 51.7 | 58.5
  Pain: Mild (n=359, 377) | 50.1 | 54.1
  Pain: Moderate (n=306, 330) | 7.5 | 23.6
  Pain: Severe (n=299, 306) | 1.3 | 2.3
  Limitation of arm movement: Any (n=313, 326) | 10.5 | 27.6
  Limitation of arm movement: Mild (n=312, 322) | 10.3 | 25.2
  Limitation of arm movement: Moderate (n=297, 303) | 0.3 | 2.6
  Limitation of arm movement: Severe (n=298, 305) | 0.7 | 3.0
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Redness: any; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -11.4, 95% CI 2-sided [-17.3 to -5.6] — Exact 2-sided confidence interval and corresponding p-value (based on Chan & Zhang) for the difference in proportions, [13vPnC] - [23vPS], expressed as a percentage
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS; Redness: mild; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.129, Chan & Zhang; difference in proportions = -4.0, 95% CI 2-sided [-9.1 to 1.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 23vPS; Redness: moderate; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.002, Chan & Zhang; difference in proportions = -6.8, 95% CI 2-sided [-11.3 to -2.3] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 23vPS; Redness: severe; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.028, Chan & Zhang; difference in proportions = -3.2, 95% CI 2-sided [-6.3 to -0.3] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 23vPS; Swelling: any; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -12.7, 95% CI 2-sided [-18.5 to -7.0] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 23vPS; Swelling: mild; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.048, Chan & Zhang; difference in proportions = -5.1, 95% CI 2-sided [-10.2 to -0.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 23vPS; Swelling: moderate; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -9.6, 95% CI 2-sided [-14.2 to -5.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 23vPS; Swelling: severe; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -4.8, 95% CI 2-sided [-7.9 to -2.7] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 23vPS; Pain: any; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.062, Chan & Zhang; Chan & Zhang = -6.8, 95% CI 2-sided [-14.0 to 0.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 23vPS; Pain: mild; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.284, Chan & Zhang; difference in proportions = -4.0, 95% CI 2-sided [-11.3 to 3.3] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 23vPS; Pain: moderate; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -16.1, 95% CI 2-sided [-21.7 to -10.6] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 23vPS; Pain: severe; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.539, Chan & Zhang; difference in proportions = -0.9, 95% CI 2-sided [-3.5 to 1.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 23vPS; Limitation of arm movement: any; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -17.1, 95% CI 2-sided [-23.1 to -11.1] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC vs 23vPS; Limitation of arm movement: mild; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p < 0.001, Chan & Zhang; difference in proportions = -14.9, 95% CI 2-sided [-20.8 to -9.0] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC vs 23vPS; Limitation of arm movement: moderate; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.020, Chan & Zhang; difference in proportions = -2.3, 95% CI 2-sided [-4.8 to -0.4] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC vs 23vPS; Limitation of arm movement: severe; difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.042, Limitation of arm movement: any; differe; difference in proportions = -2.3, 95% CI 2-sided [-4.9 to -0.1] — [estimate comment as in outcome 7, analysis 1]

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 7
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any local reaction reactogenicity events; (n)=number of participants with known values for 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 13vPnC / 13vPnC
Number analyzed (Participants) | 265 | 265
percentage of participants
  Redness: Any (n=185, 185) | 9.7 | 12.4
  Redness: Mild (n=182, 182) | 8.2 | 6.0
  Redness: Moderate (n=182, 182) | 4.4 | 7.1
  Redness: Severe (n=179, 179) | 1.1 | 1.7
  Swelling: Any (n=185, 185) | 9.2 | 10.8
  Swelling: Mild (n=182, 182) | 6.6 | 8.8
  Swelling: Moderate (n=179, 179) | 3.4 | 2.8
  Swelling: Severe (n=177, 177) | 0.0 | 0.0
  Pain: Any (n=258, 258) | 55.0 | 57.4
  Pain: Mild (n=251, 251) | 53.0 | 54.2
  Pain: Moderate (n=187, 187) | 8.6 | 11.2
  Pain: Severe (n=179, 179) | 1.7 | 0.6
  Limitation of arm movement: Any (n=195, 195) | 9.7 | 13.3
  Limitation of arm movement: Mild (n=194, 194) | 9.3 | 13.4
  Limitation of arm movement: Moderate (n=178, 178) | 0.6 | 0.6
  Limitation of arm movement: Severe (n=178, 178) | 0.6 | 0.0

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for 23vPS (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 7
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any local reaction reactogenicity events; (n)=number of participants with known values for 23vPS (Year 0) and 13vPnC / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 23vPS | 13vPnC / 13vPnC
Number analyzed (Participants) | 387 | 304
percentage of participants
  Redness: Any (n=324, 236) | 22.2 | 12.7
  Redness: Mild (n=311, 233) | 13.5 | 6.9
  Redness: Moderate (n=314, 231) | 11.5 | 6.9
  Redness: Severe (n=310, 227) | 4.8 | 1.8
  Swelling: Any (n=333, 236) | 23.1 | 12.3
  Swelling: Mild (n=315, 234) | 14.0 | 10.3
  Swelling: Moderate (n=323, 229) | 13.6 | 3.5
  Swelling: Severe (n=310, 227) | 4.8 | 0.9
  Pain: Any (n=383, 297) | 58.5 | 58.2
  Pain: Mild (n=377, 291) | 54.1 | 54.3
  Pain: Moderate (n=330, 239) | 23.6 | 13.0
  Pain: Severe (n=306, 226) | 2.3 | 0.4
  Limitation of arm movement: Any (n=326, 247) | 27.6 | 16.2
  Limitation of arm movement: Mild (n=322, 245) | 25.2 | 15.5
  Limitation of arm movement: Moderate (n=303, 228) | 2.6 | 0.9
  Limitation of arm movement: Severe (n=305, 228) | 3.0 | 0.9

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2 / Year 1 )
Description: as for outcome 7
Time Frame: Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any local reaction reactogenicity events; (n)=number of participants with known values for 13vPnC / 13vPnC and 23vPS / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Groups:
- 23vPS / 13vPnC: 23vPS 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax 2)
Arm/Group | 13vPnC / 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 304 | 311
percentage of participants
  Redness: Any (n=236, 228) | 12.7 | 10.1
  Redness: Mild (n=233, 226) | 6.9 | 8.8
  Redness: Moderate (n=231, 223) | 6.9 | 3.6
  Redness: Severe (n=227, 222) | 1.8 | 0.9
  Swelling: Any (n=236, 241) | 12.3 | 14.1
  Swelling: Mild (n=234, 236) | 10.3 | 11.9
  Swelling: Moderate (n=229, 229) | 3.5 | 4.8
  Swelling: Severe (n=227, 222) | 0.9 | 0.5
  Pain: Any (n=297, 302) | 58.2 | 56.6
  Pain: Mild (n=291, 297) | 54.3 | 53.5
  Pain: Moderate (n=239, 236) | 13.0 | 13.1
  Pain: Severe (n=226, 221) | 0.4 | 0.9
  Limitation of arm movement: Any (n=247, 251) | 16.2 | 19.9
  Limitation of arm movement: Mild (n=245, 249) | 15.5 | 18.9
  Limitation of arm movement: Moderate (n=228, 222) | 0.9 | 0.9
  Limitation of arm movement: Severe (n=228, 222) | 0.9 | 1.4

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for 13vPnC (Vax 1 / Year 0) and 23vPS / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 7
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any local reaction reactogenicity events; (n)=number of participants with known values for 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 370 | 311
percentage of participants
  Redness: Any (n=306, 228) | 10.8 | 10.1
  Redness: Mild (n=304, 226) | 9.5 | 8.8
  Redness: Moderate (n=301, 223) | 4.7 | 3.6
  Redness: Severe (n=299, 222) | 1.7 | 0.9
  Swelling: Any (n=307, 241) | 10.4 | 14.1
  Swelling: Mild (n=305, 236) | 8.9 | 11.9
  Swelling: Moderate (n=299, 229) | 4.0 | 4.8
  Swelling: Severe (n=297, 222) | 0.0 | 0.5
  Pain: Any (n=362, 302) | 51.7 | 56.6
  Pain: Mild (n=359, 297) | 50.1 | 53.5
  Pain: Moderate (n=306, 236) | 7.5 | 13.1
  Pain: Severe (n=299, 221) | 1.3 | 0.9
  Limitation of arm movement: Any (n=313, 251) | 10.5 | 19.9
  Limitation of arm movement: Mild (n=312, 249) | 10.3 | 18.9
  Limitation of arm movement: Moderate (n=297, 222) | 0.3 | 0.9
  Limitation of arm movement: Severe (n=298, 222) | 0.7 | 1.4

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for 13vPnC and 23vPS (Vax 1 / Year 0)
Description: Systemic events reported using electronic diary. Fever scaled as Any (≥38 degrees Celsius [C]); Mild (≥38 but <38.5 degrees C); Moderate (≥38.5 but <39 degrees C); Severe (≥39 but ≤40 degrees C); Potentially life-threatening (>40 degrees C). Other systemic events include Fatigue, Headache, Chills, Rash, Vomiting, Decreased appetite, New generalized muscle pain (New muscle pain), Aggravated generalized muscle pain (Aggravated muscle pain), New generalized joint pain (New joint pain), and Aggravated generalized joint pain (Aggravated joint pain).
Time Frame: Days 1 through 14 / Year 0
Population: Safety population; N=number of participants who reported any systemic reactogenicity events; (n)=number of participants with known values for 13vPnC and 23vPS (Year 0). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 388 | 403
percentage of participants
  Fever: Any ≥38 degrees C (n=299, 309) | 1.0 | 4.2
  Fever: Mild ≥38 but <38.5 degrees C (n=299, 303) | 1.0 | 2.0
  Fever: Moderate ≥38.5 but <39 degrees C(n=297,301) | 0.0 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C (n=297, 301) | 0.0 | 0.3
  Potentially life-threatening >40C (n=297, 307) | 0.0 | 2.0
  Fatigue (n=350, 367) | 34.0 | 43.3
  Headache (n=329, 331) | 23.7 | 26.0
  Chills (n=305, 312) | 7.9 | 11.2
  Rash (n=303, 323) | 7.3 | 16.4
  Vomiting (n=300, 304) | 1.7 | 1.3
  Decreased appetite (n=317, 313) | 10.4 | 11.5
  New muscle pain (n=345, 358) | 36.8 | 44.7
  Aggravated muscle pain (n=320, 334) | 20.6 | 27.5
  New joint pain (n=310, 323) | 12.6 | 14.9
  Aggravated joint pain (n=310, 322) | 11.6 | 16.5
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; New generalized muscle pain: difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.034, Chan & Zhang; difference in proportions = -7.9, 95% CI 2-sided [-15.2 to -0.6] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS; Aggravated generalized muscle pain: difference in proportions, [13vPnC] - [23vPS], expressed as a percentage; Test type: Superiority or Other; p = 0.039, Chan & Zhang; difference in proportions = -6.9, 95% CI 2-sided [-13.6 to -0.3] — [estimate comment as in outcome 7, analysis 1]

13. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 12
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any systemic reactogenicity events; (n)=number of participants with known values for 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 13vPnC / 13vPnC
Number analyzed (Participants) | 259 | 259
percentage of participants
  Fever: Any ≥38 degrees C (n=179, 179) | 1.7 | 2.2
  Fever: Mild ≥38 but <38.5 degrees C (n=179, 179) | 1.7 | 0.6
  Fever: Moderate ≥38.5 but <39 degrees C(n=177,177) | 0.0 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C (n=177, 177) | 0.0 | 0.6
  Potentially life-threatening >40C (n=177, 177) | 0.0 | 1.1
  Fatigue (n=215, 215) | 33.5 | 28.4
  Headache (n=200, 200) | 23.0 | 19.0
  Chills (n=182, 182) | 9.3 | 4.4
  Rash (n=183, 183) | 8.2 | 6.0
  Vomiting (n=178, 178) | 1.1 | 0.0
  Decreased appetite (n=190, 190) | 8.4 | 7.9
  New muscle pain (n=219, 219) | 37.9 | 35.6
  Aggravated muscle pain (n=198, 198) | 20.7 | 16.2
  New joint pain (n=187, 187) | 11.2 | 7.5
  Aggravated joint pain (n=188, 188) | 11.2 | 10.1

14. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for 23vPS (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 12
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any systemic reactogenicity events; (n)=number of participants with known values for 23vPS (Year 0) and 13vPnC / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 23vPS | 13vPnC / 13vPnC
Number analyzed (Participants) | 403 | 290
percentage of participants
  Fever: Any ≥38 degrees C (n=309, 229) | 4.2 | 3.5
  Fever: Mild ≥38 but <38.5 degrees C (n=303, 227) | 2.0 | 0.9
  Fever: Moderate ≥38.5 but <39 degrees C(n=301,227) | 0.0 | 0.9
  Fever: Severe ≥39 but ≤40 degrees C (n=301, 226) | 0.3 | 0.4
  Potentially life-threatening >40C (n=307, 227) | 2.0 | 1.3
  Fatigue (n=367, 255) | 43.3 | 28.6
  Headache (n=331, 246) | 26.0 | 19.1
  Chills (n=312, 234) | 11.2 | 7.3
  Rash (n=323, 232) | 16.4 | 6.0
  Vomiting (n=304, 226) | 1.3 | 0.4
  Decreased appetite (n=313, 237) | 11.5 | 8.9
  New muscle pain (n=358, 260) | 44.7 | 34.6
  Aggravated muscle pain (n=334, 245) | 27.5 | 18.0
  New joint pain (n=323, 238) | 14.9 | 10.5
  Aggravated joint pain (n=322, 239) | 16.5 | 12.6

15. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 12
Time Frame: Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any systemic reactogenicity events; (n)=number of participants with known values for 13vPnC / 13vPnC and 23vPS / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Groups:
- 23vPS / 13vPnC: 23vPS 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax )
Arm/Group | 13vPnC / 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 290 | 299
percentage of participants
  Fever: Any ≥38 degrees C (n=229, 224) | 3.5 | 2.2
  Fever: Mild ≥38 but <38.5 degrees C (n=227, 224) | 0.9 | 1.8
  Fever: Moderate ≥38.5 but <39 degrees C(n=227,221) | 0.9 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C (n=226, 222) | 0.4 | 0.5
  Potentially life-threatening >40C (n=227, 221) | 1.3 | 0.5
  Fatigue (n=255, 265) | 28.6 | 34.3
  Headache (n=246, 248) | 19.1 | 22.6
  Chills (n=234, 233) | 7.3 | 9.9
  Rash (n=232, 226) | 6.0 | 7.1
  Vomiting (n=226, 226) | 0.4 | 3.1
  Decreased appetite (n=237, 230) | 8.9 | 7.4
  New muscle pain (n=260, 263) | 34.6 | 35.0
  Aggravated muscle pain (n=245, 248) | 18.0 | 21.0
  New joint pain (n=238, 234) | 10.5 | 12.0
  Aggravated joint pain (n=239, 231) | 12.6 | 11.7

16. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for 13vPnC (Vax / Year 0) and 23vPS / 13vPnC (Vax 2 / Year 1)
Description: as for outcome 12
Time Frame: Days 1 through 14 / Year 0, Days 1 through 14 / Year 1
Population: Safety population; N=number of participants who reported any systemic reactogenicity events; (n)=number of participants with known values for 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 388 | 299
percentage of participants
  Fever: Any ≥38 degrees C (n=299, 224) | 1.0 | 2.2
  Fever: Mild ≥38 but <38.5 degrees C (n=299, 224) | 1.0 | 1.8
  Fever: Moderate ≥38.5 but <39 degrees C(n=297,221) | 0.0 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C (n=297, 222) | 0.0 | 0.5
  Potentially life-threatening >40C (n=297, 221) | 0.0 | 0.5
  Fatigue (n=350, 265) | 34.0 | 34.3
  Headache (n=329, 248) | 23.7 | 22.6
  Chills (n=305, 233) | 7.9 | 9.9
  Rash (n=303, 226) | 7.3 | 7.1
  Vomiting (n=300, 226) | 1.7 | 3.1
  Decreased appetite (n=317, 230) | 10.4 | 7.4
  New muscle pain (n=345, 263) | 36.8 | 35.0
  Aggravated muscle pain (n=320, 248) | 20.6 | 21.0
  New joint pain (n=310, 234) | 12.6 | 12.0
  Aggravated joint pain (n=310, 231) | 11.6 | 11.7

ADVERSE EVENTS:
Time Frame: Events assessed until approximately 1 month after each vaccination. AEs collected up to 43 days after Vax 2 / Year 1; SAEs collected up to 194 days after Vax 2 / Year 1. Local Reactions and Systemic Events assessed within 14 days of each vaccination.
Description: Same event may appear as both an AE and SAE; however, are distinct events. Event may be categorized as serious in 1 subject and nonserious in another, or 1 subject may have experienced both a serious and nonserious event during study. Zero in denominator (0 participants at risk) indicates Reporting Group was not systematically assessed for AE term.
Groups:
- 13vPnC (Vax 1 / Year 0) 1 Month After Vaccination: 13vPnC 0.5 mL dose IM at Year 0 (Vax 1)
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=66; systematic (solicited) Local Reactions N=209; systematic (solicited) Systemic Events N=234.
- 23vPS (Vax 1 / Year 0) 1 Month After Vaccination: 23vPS 0.5 mL dose IM at Year 0 (Vax 1)
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=83; systematic (solicited) Local Reactions N=248; systematic (solicited) Systemic Events N=275.
- 13vPnC 6-M FU (Vax 1 / Year 0): 13vPnC 0.5 mL dose IM at Year 0 (Vax 1); events assessed at 6-Month Follow-up visit (6-M FU) (Vax 1 / Year 0) telephone visit to report new events.
- 23vPS 6-M FU (Vax 1 / Year 0): 23vPS 0.5 mL dose IM at Year 0 (Vax 1); events assessed at 6-M FU (Vax 1 / Year 0) telephone visit to report new events.
- 13vPnC / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination: 13vPnC 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax 2)
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=69; systematic (solicited) Local Reactions N=191; systematic (solicited) Systemic Events N=161.
- 23vPS / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination: 23vPS 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax 2)
  Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=62; systematic (solicited) Local Reactions N=189; systematic (solicited) Systemic Events N=174.
- 13vPnC / 13vPnC 6-M FU (Vax 2 / Year 1): 13vPnC 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose IM at Year 1 (Vax 2) ; events assessed at 6-M FU (Vax 2 / Year 1) telephone visit to report new events.
- 23vPS / 13vPnC 6-M FU (Vax 2 / Year 1): 23vPS 0.5 mL dose IM at Year 0 (Vax 1) and 13vPnC 0.5 mL dose at Year 1 (Vax 2); events assessed at 6-M FU (Vax 2 / Year 1) telephone visit to report new events.
Arm/Group | 13vPnC (Vax 1 / Year 0) 1 Month After Vaccination | 23vPS (Vax 1 / Year 0) 1 Month After Vaccination | 13vPnC 6-M FU (Vax 1 / Year 0) | 23vPS 6-M FU (Vax 1 / Year 0) | 13vPnC / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination | 23vPS / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination | 13vPnC / 13vPnC 6-M FU (Vax 2 / Year 1) | 23vPS / 13vPnC 6-M FU (Vax 2 / Year 1)
Serious Adverse Events (participants affected / at risk) | 3/463 | 8/473 | 27/463 | 26/473 | 4/391 | 7/404 | 17/391 | 21/404
Other Adverse Events (participants affected / at risk) | 234/463 | 275/473 | 60/463 | 59/473 | 191/391 | 189/404 | 29/391 | 30/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (Vax 1 / Year 0) 1 Month After Vaccination (N=463) | 23vPS (Vax 1 / Year 0) 1 Month After Vaccination (N=473) | 13vPnC 6-M FU (Vax 1 / Year 0) (N=463) | 23vPS 6-M FU (Vax 1 / Year 0) (N=473) | 13vPnC / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination (N=391) | 23vPS / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination (N=404) | 13vPnC / 13vPnC 6-M FU (Vax 2 / Year 1) (N=391) | 23vPS / 13vPnC 6-M FU (Vax 2 / Year 1) (N=404)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3 | 4 | 1 | 0 | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC (Vax 1 / Year 0) 1 Month After Vaccination (N=463) | 23vPS (Vax 1 / Year 0) 1 Month After Vaccination (N=473) | 13vPnC 6-M FU (Vax 1 / Year 0) (N=463) | 23vPS 6-M FU (Vax 1 / Year 0) (N=473) | 13vPnC / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination (N=391) | 23vPS / 13vPnC (Vax 2 / Year 1) 1 Month After Vaccination (N=404) | 13vPnC / 13vPnC 6-M FU (Vax 2 / Year 1) (N=391) | 23vPS / 13vPnC 6-M FU (Vax 2 / Year 1) (N=404)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 1 | 4 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Injection site induration (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site movement impairment (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 3 | 3 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination site haematoma (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 6 | 0 | 0 | 3 | 7 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 1 | 3 | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Eye infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infecton (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Factured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biopsy skin (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type I diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 4 | 1 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dementia alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Senile dementia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal artery occlusion (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast calcification (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 3 | 4 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 2 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Campbell de Morgan spots (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalising (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 3 | 3 | 2 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Redness (Any) (Skin and subcutaneous tissue disorders) | 33/306 | 72/324 | 0/0 | 0/0 | 30/236 | 23/228 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 29/304 | 42/311 | 0/0 | 0/0 | 16/233 | 20/226 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 14/301 | 36/314 | 0/0 | 0/0 | 16/231 | 8/223 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 5/299 | 15/310 | 0/0 | 0/0 | 4/227 | 2/222 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 32/307 | 77/333 | 0/0 | 0/0 | 29/236 | 34/241 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 27/305 | 44/315 | 0/0 | 0/0 | 24/234 | 28/236 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 12/299 | 44/323 | 0/0 | 0/0 | 8/229 | 11/229 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/297 | 15/310 | 0/0 | 0/0 | 2/227 | 1/222 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Pain (Any) (Skin and subcutaneous tissue disorders) | 187/362 | 224/383 | 0/0 | 0/0 | 173/297 | 171/302 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 180/359 | 204/377 | 0/0 | 0/0 | 158/291 | 159/297 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 23/306 | 78/330 | 0/0 | 0/0 | 31/239 | 31/236 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 4/299 | 7/306 | 0/0 | 0/0 | 1/226 | 2/221 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 33/313 | 90/326 | 0/0 | 0/0 | 40/247 | 50/251 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 32/312 | 81/322 | 0/0 | 0/0 | 38/245 | 47/249 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 1/297 | 8/303 | 0/0 | 0/0 | 2/228 | 2/222 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 2/298 | 9/305 | 0/0 | 0/0 | 2/228 | 3/222 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Redness (Any) (Skin and subcutaneous tissue disorders) | 18/185 | 0 | 0/0 | 0/0 | 23/185 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 15/182 | 0 | 0/0 | 0/0 | 11/182 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 8/182 | 0 | 0/0 | 0/0 | 13/182 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 2/179 | 0 | 0/0 | 0/0 | 3/179 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 17/185 | 0 | 0/0 | 0/0 | 20/185 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 12/182 | 0 | 0/0 | 0/0 | 16/182 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 6/179 | 0 | 0/0 | 0/0 | 5/179 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/177 | 0 | 0/0 | 0/0 | 0/177 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Pain (Any) (Skin and subcutaneous tissue disorders) | 142/258 | 0 | 0/0 | 0/0 | 148/258 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 133/251 | 0 | 0/0 | 0/0 | 136/251 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 16/187 | 0 | 0/0 | 0/0 | 21/187 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 3/179 | 0 | 0/0 | 0/0 | 1/179 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 19/195 | 0 | 0/0 | 0/0 | 26/195 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 18/194 | 0 | 0/0 | 0/0 | 26/194 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 1/178 | 0 | 0/0 | 0/0 | 1/178 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 1/178 | 0 | 0/0 | 0/0 | 0/178 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fever (Any) ≥ 38 degrees Celsius (C) (General disorders) | 3/299 | 13/309 | 0/0 | 0/0 | 8/229 | 5/224 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fever (Mild) ≥ 38 degrees but < 38.5 degrees C (General disorders) | 3/299 | 6/303 | 0/0 | 0/0 | 2/227 | 4/224 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fever (Moderate) ≥ 38.5 degrees but < 39 degrees C (General disorders) | 0/297 | 0/301 | 0/0 | 0/0 | 2/227 | 0/221 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fever (Severe) ≥ 39 degrees but ≤ 40 degrees C (General disorders) | 0/297 | 1/301 | 0/0 | 0/0 | 1/226 | 1/222 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fever (Potentially life threatening) > 40 degrees C (General disorders) | 0/297 | 6/307 | 0/0 | 0/0 | 3/227 | 1/221 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fatigue (General disorders) | 119/350 | 159/367 | 0/0 | 0/0 | 73/255 | 91/265 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Headache (General disorders) | 78/329 | 86/331 | 0/0 | 0/0 | 47/246 | 56/248 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Chills (General disorders) | 24/305 | 35/312 | 0/0 | 0/0 | 17/234 | 23/233 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Rash (General disorders) | 22/303 | 53/323 | 0/0 | 0/0 | 14/232 | 16/226 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Vomiting (General disorders) | 5/300 | 4/304 | 0/0 | 0/0 | 1/226 | 7/226 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Decreased appetite (General disorders) | 33/317 | 36/313 | 0/0 | 0/0 | 21/237 | 17/230 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
New generalized muscle pain (General disorders) | 127/345 | 160/358 | 0/0 | 0/0 | 90/260 | 92/263 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Aggravated generalized muscle pain (General disorders) | 66/320 | 92/334 | 0/0 | 0/0 | 44/245 | 52/248 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
New generalized joint pain (General disorders) | 39/310 | 48/323 | 0/0 | 0/0 | 25/238 | 28/234 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Aggravated generalized joint pain (General disorders) | 36/310 | 53/322 | 0/0 | 0/0 | 30/239 | 27/231 | 0/0 | 0/0 — 13vPnC and 23vPS (Vax 1 / Year 0); 13vPnC / 13vPnC and 23vPS / 13vPnC (Vax 2/ Year 1)
Fever (Any) ≥ 38 degrees C (General disorders) | 3/179 | 0 | 0/0 | 0/0 | 4/179 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fever (Mild) ≥ 38 degrees but < 38.5 degrees C (General disorders) | 3/179 | 0 | 0/0 | 0/0 | 1/179 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fever (Moderate) ≥ 38.5 degrees but < 39 degrees C (General disorders) | 0/177 | 0 | 0/0 | 0/0 | 0/177 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fever (Severe) ≥ 39 degrees but ≤ 40 degrees C (General disorders) | 0/177 | 0 | 0/0 | 0/0 | 1/177 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fever (Potentially life threatening) > 40 degrees C (General disorders) | 0/177 | 0 | 0/0 | 0/0 | 2/177 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Fatigue (General disorders) | 72/215 | 0 | 0/0 | 0/0 | 61/215 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Headache (General disorders) | 46/200 | 0 | 0/0 | 0/0 | 38/200 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Chills (General disorders) | 17/182 | 0 | 0/0 | 0/0 | 8/182 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Rash (General disorders) | 15/183 | 0 | 0/0 | 0/0 | 11/183 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Vomiting (General disorders) | 2/178 | 0 | 0/0 | 0/0 | 0/178 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Decreased appetite (General disorders) | 16/190 | 0 | 0/0 | 0/0 | 15/190 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
New generalized muscle pain (General disorders) | 83/219 | 0 | 0/0 | 0/0 | 78/219 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Aggravated generalized muscle pain (General disorders) | 41/198 | 0 | 0/0 | 0/0 | 32/198 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
New generalized joint pain (General disorders) | 21/187 | 0 | 0/0 | 0/0 | 14/187 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)
Aggravated generalized joint pain (General disorders) | 21/188 | 0 | 0/0 | 0/0 | 19/188 | 0 | 0/0 | 0/0 — 13vPnC (Vax 1 / Year 0) and 13vPnC / 13vPnC (Vax 2 / Year 1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.